CLINICAL TRIAL: NCT05463289
Title: Implementing Digital Retinal Exams Into Comprehensive Pediatric Diabetes Care
Brief Title: ACCESS 2: AI for pediatriC diabetiC Eye examS Study 2
Acronym: ACCESS2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Eye Institute (NEI) (NIH); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB00180692; 1R01EY033233-01 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes; Cystic Fibrosis-related Diabetes
Keywords: Diabetic Retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetic Retinopathy

STUDY DESIGN:
Masking Description: All participants will undergo point-of-care diabetic retinopathy screening. Participants will know that they will undergo point-of-care diabetic retinopathy screening at the time of consenting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Diabetic Retinopathy Exam at the point of care (Other): Participants will undergo a point of care diabetic retinopathy eye exam using autonomous AI. Those that test positive will be referred to Eye Care Provider for dilated eye exam.
  Interventions: Diagnostic Test: Point of Care Autonomous AI diabetic retinopathy exam

INTERVENTIONS:
Diagnostic Test: Point of Care Autonomous AI diabetic retinopathy exam — Participants will undergo point-of-care diabetic retinopathy screening using autonomous artificial intelligence software to interpret retinal images taken with a non-mydriatic fundus camera and providing an immediate result.
  Other Names: IDx-DR

SUMMARY:
The purpose of this study is to determine if use of a nonmydriatic fundus camera using autonomous artificial intelligence software at the point of care increases the proportion of underserved youth with diabetes screened for diabetic retinopathy, and to determine the diagnostic accuracy of the autonomous AI system in detecting diabetic retinopathy from retinal images of youth with diabetes.

DETAILED DESCRIPTION:
This study will recruit up to 500 individuals ages 8-21 with type 1 or type 2 diabetes. In this study, participants will undergo a point-of-care diabetic eye exam using autonomous AI software on a non-mydriatic fundus camera. Participants will receive the diabetic eye exam results immediately from the autonomous AI system, and if abnormal will be referred to an eye care provider for a dilated eye exam.

In the AI for ChildrenS Diabetic Eye ExamS Study (ACCESS2), 398 participants will be enrolled to determine if point of care autonomous AI increases the proportion of minority and underserved youth screened for diabetic retinopathy. The autonomous AI interpretation will also be compared to consensus grading of retinal specialists to determine if there is agreement and to determine the diagnostic accuracy of the system in youth.

A cohort of youth with known diabetic retinopathy (true positives) will also be enrolled as an enriched population to determine the diagnostic accuracy of autonomous AI compared to the prognostic standard interpretation of a central reading center.

ELIGIBILITY:
Inclusion Criteria:

Meets American Diabetes Association (ADA) criteria for diabetic retinopathy screening:

* Diagnosis of Type 1 diabetes for ≥3 years, and age 11 or in puberty
* Diagnosis of Type 2 diabetes

Enriched cohort:

* Patients with Type 1 or Type 2 diabetes,
* 8-21 years of age with known diabetic retinopathy (true positives).
* No time limit on last diabetic eye exam.

Exclusion Criteria:

* Known diabetic eye exam in the last 12 months

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-07-11 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion screened for diabetic retinopathy | Day 1
  Equivalence in proportion screened for diabetic retinopathy of white and non-white youth with autonomous AI

SECONDARY OUTCOMES:
Percentage of agreement in interpretation of retinal images | Day 1
  Agreement in interpretation of retinal images between autonomous AI and consensus grading by ophthalmologists
Sensitivity of autonomous AI vs. prognostic standard | Day 1
  Sensitivity of autonomous AI in detecting diabetic retinopathy in youth compared to the prognostic standard. This will be analyzed in the ACCESS2 trial cohort alone, and also in the ACCESS2 trial cohort with the enriched cohort of youth with known diabetic retinopathy.
Specificity of autonomous AI vs. prognostic standard | Day 1
  Specificity of autonomous AI in detecting diabetic retinopathy in youth compared to the prognostic standard. This will be analyzed in the ACCESS2 trial cohort alone, and also in the ACCESS2 trial cohort with the enriched cohort of youth with known diabetic retinopathy.
Proportion with diabetic retinopathy | Day 1
  Proportion of participants with diabetic retinopathy, including none, mild, moderate or severe DR.

CONTACTS AND LOCATIONS:
Overall Officials: Risa M Wolf, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Pediatric Diabetes Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Channa R, Wolf R, Abramoff MD. Autonomous Artificial Intelligence in Diabetic Retinopathy: From Algorithm to Clinical Application. J Diabetes Sci Technol. 2021 May;15(3):695-698. doi: 10.1177/1932296820909900. Epub 2020 Mar 4. PMID 32126819
- [Background] Thomas CG, Channa R, Prichett L, Liu TYA, Abramoff MD, Wolf RM. Racial/Ethnic Disparities and Barriers to Diabetic Retinopathy Screening in Youths. JAMA Ophthalmol. 2021 Jul 1;139(7):791-795. doi: 10.1001/jamaophthalmol.2021.1551. PMID 34042939
- [Background] Wolf RM, Channa R, Abramoff MD, Lehmann HP. Cost-effectiveness of Autonomous Point-of-Care Diabetic Retinopathy Screening for Pediatric Patients With Diabetes. JAMA Ophthalmol. 2020 Oct 1;138(10):1063-1069. doi: 10.1001/jamaophthalmol.2020.3190. PMID 32880616
- [Background] Wolf RM, Liu TYA, Thomas C, Prichett L, Zimmer-Galler I, Smith K, Abramoff MD, Channa R. The SEE Study: Safety, Efficacy, and Equity of Implementing Autonomous Artificial Intelligence for Diagnosing Diabetic Retinopathy in Youth. Diabetes Care. 2021 Mar;44(3):781-787. doi: 10.2337/dc20-1671. Epub 2021 Jan 21. PMID 33479160
- [Background] Porter M, Channa R, Wagner J, Prichett L, Liu TYA, Wolf RM. Prevalence of diabetic retinopathy in children and adolescents at an urban tertiary eye care center. Pediatr Diabetes. 2020 Aug;21(5):856-862. doi: 10.1111/pedi.13037. Epub 2020 May 31. PMID 32410329